CLINICAL TRIAL: NCT05663580
Title: Cohort Study of HIV-positive People, Treated With Long Acting Antiretroviral Therapy (SCohoLART)
Brief Title: Cohort Study of HIV-positive People, Treated With Long Acting Antiretroviral Therapy
Acronym: SCohoLART
Status: Recruiting | Type: Observational
Sponsor: Castagna Antonella (Other)
Responsible Party: Sponsor-Investigator, Castagna Antonella, Professor, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: v1.0, 18-03-2022
Record Dates: First submitted 2022-11-21; First posted 2022-12-23 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections
Keywords: HIV therapy; PLWH; long-acting antiretroviral drugs; cabotegravir; rilpivirine
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Rilpivirine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HIV-positive people virologically suppressed without resistance/failure to NNRTI and INI: Initial administration of two separate intramuscolar injection of cabotegravir 400mg/3mL and rilpivirine 600mg/3mL in opposite gluteal muscles, repeated one month later and then every two months.
  Interventions: Drug: Cabotegravir 600mg/3mL, Rilpivirine 900mg/3mL

INTERVENTIONS:
Drug: Cabotegravir 600mg/3mL, Rilpivirine 900mg/3mL — Initial administration of two separate intramuscolar injection of cabotegravir 400mg/3mL and rilpivirine 600mg/3mL in opposite gluteal muscles, repeated one month later and then every two months.

SUMMARY:
Systematic, continuative collection of clinical and laboratory data on patients followed at lnfectious Diseases Unit of the IRCCS San Raffaele Hospital in Milan, receiving long-acting ART (Phase IV, single-center, prospective, cohort study)

PRIMARY ENDOPOINT: Treatment failure over 48 weeks, defined as virological failure (VF) or therapy discontinuation for any reason (TD)

SECONDARY ENDPOINTS:

Clinical and pharmacological determinants of efficacy, tolerability, toxicity Modifications in risk and incidence of comorbidities Description of drug-resistance in case of VR Efficacy of rescue regimens in case of VF Quality of life and patient's satisfaction

DETAILED DESCRIPTION:
The SCohoLART Study consists of the systematic, continuative collection of clinical and laboratory data on patients followed at the Centro San Luigi (lnfectious Diseases) of the IRCCS Ospedale San Raffaele in Milano, receiving long-acting ART regimens.

Currently the Centro San Luigi follows-up·5122 HIV-infected patients; we hypothesize that at least one third of them (roughly 1500) could be initially eligible for a long-acting ART with cabotegravir and rilpivirine

The collection of study related clinical and laboratory information, as well as study specific blood samples, will start only after the patient has given and dated/signed his/her informed consent to participate in the study.

Patients enrolled in this cohort will be followed according to the standard of care; they will receive the prescribed long-acting regimen according to the indication and posology authorized by AIFA and described in the technical sheet of the drug(s). Follow-up ambulatory visits and laboratory tests will be generally performed every 6 months (earlier, if necessary, on patient's demand or physician's opinion). According to EACS guidelines, patients with obesity, metabolic syndrome or persistent ALT elevation will be evaluated for suspected non-alcoholic fatty liver disease (NAFLD) by ultrasonography and then by liver transient elastography (fibroscan), if NAFLD suggested by ultrasonography.

The following information will be checked and recorded at baseline:

* HIV viral load, CD4+ cell count, co-infection with viruses causing hepatitis (in particular HBV), history of AIDS-defining events;
* Smoking habit, alcohol consumption;
* Current comorbidity (including cancers, diabetes, cardio-vascular, kidney and liver diseases, psychiatric disorders (with focus on depression), sexually transmitted diseases;
* concomitant medications;
* lipid profile, glycemic metabolisms;
* if previously performed, results of drug resistance testing.

The following information will be acquired at each follow-up visit:

* general clinical evaluation (e.g. symptoms, new clinical events, including adverse events, vital signs);
* results of the last routine laboratory tests;
* results of other investigations (e.g. radiological evaluations, ultrasonography);
* concomitant medications;
* Abdominal circumference and weight;
* Systolic and diastolic blood pressure;
* Drug plasma concentrations;
* lnterval since last injection;
* Quality of life and patient's satisfaction.

Adjunctive blood samples (28 ml) will be collected and then stored at the following timepoints:

* Baseline (start of the long-acting regimen)
* Every 1 year thereafter or at the stop the long-acting regimen.

Investigations that will be performed on stored blood samples are not fully anticipated; they will be gradually defined in consequence of clinical issues that will emerge during patients' follow-up. It can be anticipated that these investigations will include biomarkers of central nervous system toxicity and of HBV monitoring in patients who are HBsAg-negative, but HBcAb-positive.

The study is observational; if necessary, the antiretroviral therapy will be modified by the reference physician, according to the standard of care; the participation in the protocol will not influence any therapeutic decision.

Adverse events will be managed according to the post-marketing legislation: it is responsibility of the promoter/investigator to notify (as normai clinical practice) any adverse reaction occurring during the study according to the norm issued by AIFA on 20/03/2008, which applies to any adverse reaction observed by doctors or other healthcare professional, on the basis of the Decreto Ministeriale del DM issued on 30/04/2015 and following updates.

In parallel, the investigator will also notify the person in charge of the pharmacovigilance of Ospedale San Raffaele (the Director of the hospital pharmacy), by completing the adverse reaction form within two days from being aware of the reaction or within 36 hours if the reaction follows the administration of biological drugs, including vaccines.

The cumulative probabilities of treatment failure or virological failure or discontinuation at 12, 24, 48 weeks since the start of the study regimen will be estimated overall and according to a number of baseline characteristics by the Kaplan-Meier curve and compared by the log-rank test. These analyses will consider as baseline the date of start of the long-acting ART regimen with cabotegravir and rilpivirine; follow-up will accrue from the baseline date to the date of treatment failure/virological failure/discontinuation or last available visit.

Univariate and multivariate Cox proportional hazard regression models will be performed to identify baseline factors associated with treatment failure. Baseline covariates with a statistically significant (p<0.05) or marginally significant (p-value <0.20) difference between people with or without treatment failure at univariate analyses and other baseline characteristics known to be associated with the study outcome will be entered into the multivariate model. Variables will be assessed for multicollinearity before inclusion into the final multivariate model.

The analysis will also assess significant changes in laboratory parameters occurred during the treatment with the study regimen by univariate mixed linear models (with random slope and random intercept), if more than 2 determinations will be available during the considered follow-up; otherwise absolute changes between the baseline and last available determination (untimed) will be calculated and tested by the Wilcoxon signed-rank test.

The analyses will be conducted using two-sided test at 0.05 alpha level of significance and using SAS v 9.4 (Cary, NC).

Data will be collected and filed by means of the electronic clinical chart for ambulatory patients currently in use at the Centro San Luigi (Malattie Infettive), IRCCS Ospedale San Raffaele in Milano for the routine management of HIV-infected patients followed at the aforementioned center.

All data extracted from patient charts will be de-identified. Only the investigators, and the clinical staff involved in this study, will have access to the de-identified data. All data will be protected from unauthorized access. The data will be stored and recorded in an electronic database in pseudo-anonymous form. The details of the names or initials will be replaced by a number and/or an alphabetic code, possibly with the year of birth of the patients. All documents will be stored in a protected place.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection;
* Age > 18 years;
* HIV-RNA <50 copies/ml;
* Stable ART;
* Planned start of a long-acting regimen approved by AIFA (initially, cabotegravir and rilpivirine);
* Written informed consent provided.

Exclusion Criteria:

- Any contraindication to the use of one or more long-acting drug, according to the technical sheet of the long-acting drug(s) planned to be started (including pregnancy, current or planned).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include HIV-infected patients, followed at IRCCS Ospedale San Raffaele in Milano, who are virologically suppressed (HIV-1 RNA <50 copies/mL) on a stable antiretroviral regimen without present or past evidence of viral resistance to, and no prior virological failure with agents of the NNRTI and INI class.
  Patients will be included in the cohort only after having agreed with the reference physician to switch from the current to a long-acting ART regimen, only after AIFA has approved the long-acting regimen planned to be started, and only after having given their informed consent to participate in the cohort and to have their anonymized clinical and laboratory data analyzed for scientific purpose.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-07-17 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2027-07-17 (Estimated)

PRIMARY OUTCOMES:
Cumulative proportion of people with treatment failure | 48 weeks
  The primary study endpoint will be the cumulative proportion of people with treatment failure over 48 weeks. Treatment failure is defined by the occurrence of virological failure (2 consecutive HIV-RNA values >50 copies/mL or a single HIV-RNA value >1000 copies/mL after the start of a long-acting ART with cabotegravir and rilpivirine) or discontinuation for any reason of the study regimen.
  The SCohoLART Study wants to collect clinical data on HIV-infected patients treated with long-acting regimens approved by AIFA (cabotegravir and rilpivirina), in order to optimize during a long-term follow-up their clinical management.

SECONDARY OUTCOMES:
Cumulative proportion of people with experience of toxic effects | 48 weeks
  The secondary outcome is the cumulative proportion of people who experience toxic effects in order to define tolerability and toxicity (including reasons for stopping).
Cumulative proportion of individuals with HIV-RNA <50 copies/mL at 1 and 2 years | 48 weeks
  As secondary outcome we want to define clinical and pharmacological determinants of efficacy at 1 and 2 years
Triglycerides (mg/dl) as values of risk comorbidities | 48 weeks
  As secondary outcome we want to describe possible modifications in the risk of comorbidities (including BMI, lipid profile, renal function and liver fibrosis)
Total cholesterol (mg/dl) as values of risk comorbidities | 48 weeks
  As secondary outcome we want to describe possible modifications in the risk of comorbidities (including BMI, lipid profile, renal function and liver fibrosis)
High density lipoprotein cholesterol (HDL, mg/dl) as values of risk comorbidities | 48 weeks
  As secondary outcome we want to describe possible modifications in the risk of comorbidities (including BMI, lipid profile, renal function and liver fibrosis)
Low density lipoprotein cholesterol (LDL, mg/dl) as values of risk comorbidities | 48 weeks
  As secondary outcome we want to describe possible modifications in the risk of comorbidities (including BMI, lipid profile, renal function and liver fibrosis)
Creatinine (mg/dl) as values of risk comorbidities | 48 weeks
  As secondary outcome we want to describe possible modifications in the risk of comorbidities (including BMI, lipid profile, renal function and liver fibrosis)
Glucose (mg/dl) as values of risk comorbidities | 48 weeks
  As secondary outcome we want to describe possible modifications in the risk of comorbidities (including BMI, lipid profile, renal function and liver fibrosis)
BMI (kg/m^2) as values of risk comorbidities | 48 weeks
  As secondary outcome we want to describe possible modifications in the risk of comorbidities (including weight in kilograms, BMI, lipid profile and changes in fat accumulation in the liver)
Incidence of new comorbidities | 48 weeks
  Incidence of new comorbidities
Cumulative proportion and features of drug-resistance | 48 weeks
  Description of drug-resistance in case of virological failure
Proportion of individuals achieving virological success (HIV-RNA <50 copies/mL) with new ART regimens in case of virological failure | 48 weeks
  Efficacy of rescue regimens in case of virological failure
w-bq12 questionnaire | 48 weeks
  Quality of life and patient's satisfaction

OTHER OUTCOMES:
Proportion of people with treatment failure and time to treatment failure | 5 years
  Cumulative proportion of people with treatment failure over 2, 3, 4 and 5 years since the start of the study regime and time to treatment failure, including estimates of cumulative probabilities of treatment failure at 12, 24, 48 weeks, at 2, 3, 4 and 5 years since the start of the study regimen.
Potential clinical and pharmacological predictors of risk of treatment failure | 48 weeks
  Risk of treatment failure according to a number of potential clinical and pharmacological predictors at 12, 24, 48 weeks
Cumulative proportion of people with virological failure | 5 years
  Proportion of people with virological failure at 1, 2, 3, 4 and 5 years
Time to virological failure | 5 years
  Time to virological failure, including estimates of probabilities of virological failure at 12, 24, 48 weeks, at 2, 3, 4 and 5 years
Cumulative proportion of therapy discontinuation | 5 years
  Proportion of patients who discontinued the study regimen for any reason, frequency of the reason leading to discontinuation and time to discontinuation over 48 weeks and over 2, 3, 4 and 5 years
Incidence of new comorbidities | 5 years
  Incidence of new comorbidities over 48 weeks and over 2, 3, 4 and 5 years
Frequency of new drug resistant variants | 5 years
  Frequency of new drug resistant variants in case of virological failure
Cumulative proportion of virological success with new ART regimens | 5 years
  Proportion of individuals achieving virological success (HIV-RNA <50 copies/mL) with new ART regimens in case of virological failure with a long-acting ART with cabotegravir and rilpivirine

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele Scientific Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Margolis DA, Gonzalez-Garcia J, Stellbrink HJ, Eron JJ, Yazdanpanah Y, Podzamczer D, Lutz T, Angel JB, Richmond GJ, Clotet B, Gutierrez F, Sloan L, Clair MS, Murray M, Ford SL, Mrus J, Patel P, Crauwels H, Griffith SK, Sutton KC, Dorey D, Smith KY, Williams PE, Spreen WR. Long-acting intramuscular cabotegravir and rilpivirine in adults with HIV-1 infection (LATTE-2): 96-week results of a randomised, open-label, phase 2b, non-inferiority trial. Lancet. 2017 Sep 23;390(10101):1499-1510. doi: 10.1016/S0140-6736(17)31917-7. Epub 2017 Jul 24. PMID 28750935
- [Background] Jaeger H, Overton ET, Richmond G, Rizzardini G, Andrade-Villanueva JF, Mngqibisa R, Hermida AO, Thalme A, Belonosova E, Ajana F, Benn PD, Wang Y, Hudson KJ, Espanol CM, Ford SL, Crauwels H, Margolis DA, Talarico CL, Smith KY, van Eygen V, Van Solingen-Ristea R, Vanveggel S, Spreen WR. Long-acting cabotegravir and rilpivirine dosed every 2 months in adults with HIV-1 infection (ATLAS-2M), 96-week results: a randomised, multicentre, open-label, phase 3b, non-inferiority study. Lancet HIV. 2021 Nov;8(11):e679-e689. doi: 10.1016/S2352-3018(21)00185-5. Epub 2021 Oct 11. PMID 34648734
- [Background] Swindells S, Andrade-Villanueva JF, Richmond GJ, Rizzardini G, Baumgarten A, Masia M, Latiff G, Pokrovsky V, Bredeek F, Smith G, Cahn P, Kim YS, Ford SL, Talarico CL, Patel P, Chounta V, Crauwels H, Parys W, Vanveggel S, Mrus J, Huang J, Harrington CM, Hudson KJ, Margolis DA, Smith KY, Williams PE, Spreen WR. Long-Acting Cabotegravir and Rilpivirine for Maintenance of HIV-1 Suppression. N Engl J Med. 2020 Mar 19;382(12):1112-1123. doi: 10.1056/NEJMoa1904398. Epub 2020 Mar 4. PMID 32130809
- [Background] Overton ET, Richmond G, Rizzardini G, Jaeger H, Orrell C, Nagimova F, Bredeek F, Garcia Deltoro M, Swindells S, Andrade-Villanueva JF, Wong A, Khuong-Josses MA, Van Solingen-Ristea R, van Eygen V, Crauwels H, Ford S, Talarico C, Benn P, Wang Y, Hudson KJ, Chounta V, Cutrell A, Patel P, Shaefer M, Margolis DA, Smith KY, Vanveggel S, Spreen W. Long-acting cabotegravir and rilpivirine dosed every 2 months in adults with HIV-1 infection (ATLAS-2M), 48-week results: a randomised, multicentre, open-label, phase 3b, non-inferiority study. Lancet. 2021 Dec 19;396(10267):1994-2005. doi: 10.1016/S0140-6736(20)32666-0. Epub 2020 Dec 9. PMID 33308425
- [Background] Rizzardini G, Overton ET, Orkin C, Swindells S, Arasteh K, Gorgolas Hernandez-Mora M, Pokrovsky V, Girard PM, Oka S, Andrade-Villanueva JF, Richmond GJ, Baumgarten A, Masia M, Latiff G, Griffith S, Harrington CM, Hudson KJ, St Clair M, Talarico CL, Patel P, Cutrell A, Van Eygen V, D'Amico R, Mrus JM, Wu S, Ford SL, Chow K, Roberts J, Wills A, Walters N, Vanveggel S, Van Solingen-Ristea R, Crauwels H, Smith KY, Spreen WR, Margolis DA. Long-Acting Injectable Cabotegravir + Rilpivirine for HIV Maintenance Therapy: Week 48 Pooled Analysis of Phase 3 ATLAS and FLAIR Trials. J Acquir Immune Defic Syndr. 2020 Dec 1;85(4):498-506. doi: 10.1097/QAI.0000000000002466. PMID 33136751
- [Background] Orkin C, Arasteh K, Gorgolas Hernandez-Mora M, Pokrovsky V, Overton ET, Girard PM, Oka S, Walmsley S, Bettacchi C, Brinson C, Philibert P, Lombaard J, St Clair M, Crauwels H, Ford SL, Patel P, Chounta V, D'Amico R, Vanveggel S, Dorey D, Cutrell A, Griffith S, Margolis DA, Williams PE, Parys W, Smith KY, Spreen WR. Long-Acting Cabotegravir and Rilpivirine after Oral Induction for HIV-1 Infection. N Engl J Med. 2020 Mar 19;382(12):1124-1135. doi: 10.1056/NEJMoa1909512. Epub 2020 Mar 4. PMID 32130806
- [Background] Orkin C, Bernal Morell E, Tan DHS, Katner H, Stellbrink HJ, Belonosova E, DeMoor R, Griffith S, Thiagarajah S, Van Solingen-Ristea R, Ford SL, Crauwels H, Patel P, Cutrell A, Smith KY, Vandermeulen K, Birmingham E, St Clair M, Spreen WR, D'Amico R. Initiation of long-acting cabotegravir plus rilpivirine as direct-to-injection or with an oral lead-in in adults with HIV-1 infection: week 124 results of the open-label phase 3 FLAIR study. Lancet HIV. 2021 Nov;8(11):e668-e678. doi: 10.1016/S2352-3018(21)00184-3. Epub 2021 Oct 14. PMID 34656207
- [Background] Cutrell AG, Schapiro JM, Perno CF, Kuritzkes DR, Quercia R, Patel P, Polli JW, Dorey D, Wang Y, Wu S, Van Eygen V, Crauwels H, Ford SL, Baker M, Talarico CL, Clair MS, Jeffrey J, White CT, Vanveggel S, Vandermeulen K, Margolis DA, Aboud M, Spreen WR, van Lunzen J. Exploring predictors of HIV-1 virologic failure to long-acting cabotegravir and rilpivirine: a multivariable analysis. AIDS. 2021 Jul 15;35(9):1333-1342. doi: 10.1097/QAD.0000000000002883. PMID 33730748
- [Background] Hemelaar J, Elangovan R, Yun J, Dickson-Tetteh L, Kirtley S, Gouws-Williams E, Ghys PD; WHO-UNAIDS Network for HIV Isolation and Characterisation. Global and regional epidemiology of HIV-1 recombinants in 1990-2015: a systematic review and global survey. Lancet HIV. 2020 Nov;7(11):e772-e781. doi: 10.1016/S2352-3018(20)30252-6. PMID 33128904
- [Background] Schlosser M, Kartashev VV, Mikkola VH, Shemshura A, Saukhat S, Kolpakov D, Suladze A, Tverdokhlebova T, Hutt K, Heger E, Knops E, Bohm M, Di Cristanziano V, Kaiser R, Sonnerborg A, Zazzi M, Bobkova M, Sierra S. HIV-1 Sub-Subtype A6: Settings for Normalised Identification and Molecular Epidemiology in the Southern Federal District, Russia. Viruses. 2020 Apr 22;12(4):475. doi: 10.3390/v12040475. PMID 32331438
- [Background] Charpentier C, Storto A, Soulie C, Ferre VM, Wirden M, Joly V, Lambert-Niclot S, Palich R, Morand-Joubert L, Landman R, Lacombe K, Katlama C, Ghosn J, Marcelin AG, Calvez V, Descamps D. Prevalence of genotypic baseline risk factors for cabotegravir + rilpivirine failure among ARV-naive patients. J Antimicrob Chemother. 2021 Oct 11;76(11):2983-2987. doi: 10.1093/jac/dkab161. PMID 34015097
- [Background] Wensing AM, Calvez V, Ceccherini-Silberstein F, Charpentier C, Gunthard HF, Paredes R, Shafer RW, Richman DD. 2019 update of the drug resistance mutations in HIV-1. Top Antivir Med. 2019 Sep;27(3):111-121. PMID 31634862
- [Background] Lai A, Franzetti M, Bergna A, Saladini F, Bruzzone B, Di Giambenedetto S, Di Biagio A, Lo Caputo S, Santoro MM, Maggiolo F, Parisi SG, Rusconi S, Gianotti N, Balotta C. Marked decrease in acquired resistance to antiretrovirals in latest years in Italy. Clin Microbiol Infect. 2021 Jul;27(7):1038.e1-1038.e6. doi: 10.1016/j.cmi.2020.09.028. Epub 2020 Sep 23. PMID 32979570
- [Background] Flexner C, Owen A, Siccardi M, Swindells S. Long-acting drugs and formulations for the treatment and prevention of HIV infection. Int J Antimicrob Agents. 2021 Jan;57(1):106220. doi: 10.1016/j.ijantimicag.2020.106220. Epub 2020 Nov 6. PMID 33166693
- See also: REKAMYS — https://www.ema.europa.eu/en/medicines/human/EPAR/rekambys
- See also: VOCABRIA — https://www.ema.europa.eu/en/medicines/human/EPAR/vocabria
- See also: EACS SOCIETY — http://www.eacsociety.org